CLINICAL TRIAL: NCT00259766
Title: Symbicort and Health Economics in a Real Life Evaluation - SHARE - A Randomised, Open-Label, Parallel-Group, Multicentre Study to Assess the Asthma-Related Health-Care Costs, in Ordinary Clinical Practice During 12 Months
Brief Title: SHARE - Symbicort and Health Economics in a Real Life Evaluation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5890L00001; SHARE
Record Dates: First submitted 2005-11-25; First posted 2005-12-01 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide; Budesonide, Formoterol Fumarate Drug Combination; Formoterol Fumarate; Terbutaline

INTERVENTIONS:
Drug: Budesonide
  Other Names: Symbicort
Drug: Formoterol
Drug: Terbutaline

SUMMARY:
The purpose of this study is to compare health-related costs and asthma control in ordinary clinical practice during 12 months for Symbicort® given as a low maintenance dose plus as needed compared to a free combination of Pulmicortâ and Oxis® plus Bricanyl® as needed, and Symbicort fixed dosing plus Bricanyl as needed in asthmatic patients not adequately controlled on inhaled glucocorticosteroids alone.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent,
* asthma,
* previously treated with glucocorticosteroids and B2-agonist

Exclusion Criteria:

* History of smoking, pregnancy, any significant disease or disorder which may put the patient at risk because of study participation

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1970
Dates: Start 2004-04; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Asthma-related health-care utilization as measured by total amount of asthma medication purchased and number of contacts with health-care facilities

SECONDARY OUTCOMES:
Number of days patients or assistant persons are absent from work due to patient's asthma
Number of exacerbations and treatment failures

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Symbicort Medical Science Director, MD, Study Director — AstraZeneca
Locations (108):
- Sweden (108):
  - Research Site, Alingsås
  - Research Site, Angered
  - Research Site, Arlöv
  - Research Site, Arvidsjaur
  - Research Site, Arvika
  - Research Site, Ängelholm
  - Research Site, Åkersberga
  - Research Site, Ånge
  - Research Site, Årsta
  - Research Site, Åstorp
  - Research Site, Åtvidaberg
  - Research Site, Bandhagen
  - Research Site, Boden
  - Research Site, Borensberg
  - Research Site, Bro
  - Research Site, Brunflo
  - Research Site, Eskilstuna
  - Research Site, Falun
  - Research Site, Filipstad
  - Research Site, Fränsta
  - Research Site, Gagnef
  - Research Site, Gärsnäs
  - Research Site, Gothenburg
  - Research Site, Grängesberg
  - Research Site, Gullspång
  - Research Site, Halmstad
  - Research Site, Håby
  - Research Site, Helsingborg
  - Research Site, Hisingsbacka
  - Research Site, Hofors
  - Research Site, Höganäs
  - Research Site, Höllviken
  - Research Site, Huddinge
  - Research Site, Iggesund
  - Research Site, Jarfalla
  - Research Site, Kalmar
  - Research site, Karlskoga
  - Research Site, Karlstad
  - Research Site, Katrineholm
  - Research Site, Kil
  - Research Site, Kinna
  - Research Site, Klippan
  - Research Site, Kolmården
  - Research Site, Kristinehamn
  - Research Site, Kungälv
  - Research Site, Kungsbacka
  - Research Site, Kungsör
  - Research Site, Landskrona
  - Research Site, Laxå
  - Research Site, Leksand
  - Research Site, Lerum
  - Research Site, Lidingö
  - Research Site, Likenäs
  - Research Site, Limhamn
  - Research Site, Lindome
  - Research Site, Linköping
  - Research Site, Ljungskile
  - Research Site, Ludvika
  - Research Site, Luleå
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Mariefred
  - Research Site, Mölndal
  - Research site, Mölnlycke
  - Research Site, Nacka
  - Research Site, Norrköping
  - Research Site, Norrtälje
  - Research Site, Nyköping
  - Research site, Osby
  - Research site, Ödeshög
  - Research Site, Örebro
  - Research Site, Partille
  - Research Site, Påarp
  - Reseearch Site, Perstorp
  - Research Site, Saltsjo-Bo
  - Research Site, Sandviken
  - Research Site, Sjöbo
  - Research Site, Sjuntorp
  - Research site, Sollentuna
  - Research Site, Solna
  - Research Site, Söderköping
  - Research site, Stenstorp
  - Research Site, Stenungsund
  - Research Site, Stockholm
  - Research Site, Storfors
  - Research Site, Stugun
  - Research Site, Sundbyberg
  - Research Site, Sundsvall
  - Research Site, Sunne
  - Research Site, Täby
  - Research Site, Trollhättan
  - Research Site, Trosa
  - Research Site, Tyresö
  - Research Site, Uddevalla
  - Research site, Ulricehamn
  - Research Site, Umeå
  - Research Site, Uppsala
  - Research Site, Vallentuna
  - Research Site, Varberg
  - Research Site, Vännäs
  - Research Site, Värnamo
  - Research site, Väsby
  - Research Site, Västerås
  - Research Site, Västervik
  - Research site, Västra Frölunda
  - Research Site, Vellinge
  - Research Site, Ystad
  - Research Site, Ytterby